CLINICAL TRIAL: NCT04797702
Title: A Open-label, Multi-center Phase Ib/II Clinical Study of Glumetinib Combined With Toripalimab in Patients With Relapsed or Metastatic Non-small Cell Lung Cancer Who Have Failed or Are Intolerant to Standard Therapy.
Brief Title: Glumetinib Combined With Toripalimab in the Treatment of Relapsed or Metastatic Non-small Cell Lung Cancer.
Acronym: CT32
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JS001-032-Ib/II-NSCLC
Record Dates: First submitted 2021-02-26; First posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-02

CONDITIONS: Relapsed or Metastatic Non-small Cell Lung Cancer
MeSH Terms: conditions — Recurrence; Carcinoma, Non-Small-Cell Lung | interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Glumetinib combined with Toripalimab
  Interventions: Combination Product: Glumetinib combined with Toripalimab

INTERVENTIONS:
Combination Product: Glumetinib combined with Toripalimab — Ib：All enrolled subjects received Glumetinib combined with Toripalimab on a 21-day cycle, starting with 200mg/ day continuous Glumetinib and 240mg/ 3 weeks Toripalimab.
  II：The SMC will determine the dose group for the Phase II study based on the safety and initial efficacy data of the Phase Ib subjects. Approximately 62 evaluable subjects will be enrolled in the study to receive the recommended dose of Glumetinib once daily and continuous treatment with Toripalimab 240mg every 3 weeks.

SUMMARY:
This is an open-label, multicenter Phase Ib/II registration clinical study, consisting of two parts: the Phase Ib dose-climbing study and the Phase II efficacy exploration study.

Phase Ib :

Phase Ib is a multicenter, single-arm study evaluating the safety, tolerability, and preliminary efficacy of SCC244 combined with Toripalimab in patients with advanced relapsed or metastatic non-small cell lung cancer who have failed standard therapy.At the start of the study, MTPI2 was used to guide toxicity monitoring and dose climbing in combination with Toripalimab (240mg intravenous every 3 weeks), with 5 subjects planned to be enrolled in each dose group.The SMC will decide whether to add the new dose level and sample size based on the latest study data available.The MTD or recommended phase II dose (RP2D) will be determined during the phase Ib study on the basis of the latest availablestudy data, and the phase II study will commence once the MTD or recommended phase II dose (RP2D) is confirmed.

Phase II:

Phase II is a multicenter, open-label, single-arm study evaluating the efficacy and safety of a recommended dose of glumetinib combined with Toripalimab in patients with relapsed, metastatic non-small cell lung cancer who have failed standard therapy.The SMC determined the dose group for the Phase II study based on the safety and initial efficacy data of the Phase Ib subjects.Approximately 62 evaluable subjects will be enrolled, with the recommended dose of glutmetinib once daily and Toripalimab 240mg every 3 weeks.

Every 21 days is a treatment cycle until the subject develops disease progression,intolerable toxicity, has used JS001 for 2 years, the informed consent is withdrawn, the investigator considers that the subject should not continue the medication, lost to follow-up, death occurs, or the study is terminated, whichever comes first.

ELIGIBILITY:
Inclusion criteria:

1. Subsubjects with histologically or cytologically confirmed NSCLC, clinically diagnosed as locally advanced (stage IIIB or IIIC) and stage IV NSCLC (according to AJCC 8th edition staging), EGFR wild-type, negative for ALK and ROS1 rearrangement, and no Met exon14 skipping mutation; genetic testing is not mandatory for subjects with squamous cell cancer;
2. PD - L1 expression of 1% or higher.
3. Non-small cell lung cancer patients following failure of or were intolerance to previous standard treatment (chemotherapy and immunotherapy alone or in combination) and received no more than third-line treatment;
4. At least 1 measurable tumor lesion according to RECIST1.1 criteria.
5. Subjects must provide valid and qualified tissue samples (fresh biopsy or preserved tumor tissue samples are acceptable, but fresh biopsy samples are preferred).
6. ECOG score ≤1 point;
7. Sufficient function of bone marrow, liver and kidney organs.

Exclusion criteria:

1. Pathological diagnosis confirmed the presence of small cell lung cancer;
2. The patient was currently participating in and receiving other studies or had previously received another c-Met inhibitor;
3. There are mutations/rearrangements of EGFR, ALK, ROS1, Met14 exon skipping;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2021-04-15 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2024-02-26 (Estimated)

PRIMARY OUTCOMES:
The type, frequency, severity and outcome of adverse events (TEAE) and serious adverse events (SAE) that occurred during the treatment period. (Phase Ib) | 2 years
  The toxicity was evaluated according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) (version 5.0) Grade.
Number of prticipants with abnormal laboratory values and/or Adverse Events that are related to treatment. (Phase Ib) | 2 years
  Laboratory values include 1. Routine blood test: Including complete blood count with differential. 2.Routine urine test: including specific gravity, pH, urine glucose, protein, ketone bodies and blood cell. 3.Serum biochemistry: Including ALT, AST, ALP, TP, ALB, TBIL, DBIL, GLU, BUN/UREA, Cr, K+, Na+, Cl-, Ca2+, P, TG, TC, HDL, LDL, and AMY/LIP. 4.Coagulation function: Including at least international normalized ratio (INR), activated partial thromboplastin time (APTT), fibrinogen (FIB), thrombin time (TT); if the international normalized ratio (INR) is not available, replace it with prothrombin time (PT). 5.Thyroid function test includes: serum thyroid stimulating hormone (TSH), free triiodothyronine (FT3), and free thyroxine (FT4); if FT3 and FT4 are not available, replace them with T3 and T4. 6.Troponin I or troponin T content: only during the screening period and when clinical indications (such as cardiac events occur).
Number of participants with abnormal vital signs values and/or Adverse Events that are related to treatment. (Phase Ib) | 2 years
  The vital signs include body temperature, heart rate, and respiratory frequency and blood pressure.
Number of participants with abnormal ECG and echocardiography values /or Adverse Events that are related to treatment. (Phase Ib) | 2 years
  During the screening period, it is necessary to repeat the inspection three times before the first administration, with an interval of about 5 minutes between each time. Calculate the QTc interval and calculate the mean (corrected using Fridericia's formula). If the inspection time in the screening period is ≤ 7 days before the first administration, the review may not be necessary according to the judgment of the investigator. Check once a week in the 1st cycle of phase Ib, check once on the 1st and 15th days of the 2nd cycle, and check once every 3 weeks from the 3rd cycle. Use echocardiography or multi-gate angiography scan to check the left ventricular ejection fraction.
Number of participants with aphysical examination values /or Adverse Events that are related to treatment.(Phase Ib) | 2 years
  A full physical examination in the screening period and at the end-of-treatment visit, including head, eyes, ears, nose, throat, neck, heart, chest (including lungs), abdomen, four limbs, skin, lymph nodes, nervous system, and subject's general condition. Body height and body weight are measured at the first visit, and then body weight is measured at each of the subsequent visits. Targeted physical examination will be conducted at other visits by the investigator.
To determine the recommended dose for the phase II study (RP2D) .(Phase Ib) | 2 years
  Phase Ib is the dose-escalation period, and the optimal dose of Glumetinib combined with Toripalimab was explored as the recommended dose for the phase II clinical study.
Investigator-assessed objective response rate (ORR) (Phase 2) | 2 years
  ORR refers to the percentage of subjects with confirmed CR or PR according to RECIST1.1

SECONDARY OUTCOMES:
Investigator-assessed objective response rate (ORR). (Phase 1b) | 2 years
  ORR refers to the percentage of subjects with confirmed CR or PR according to RECIST1.1 and iRECIST.
Investigator-assessed progression-free survival (PFS) . (Phase 1b) | 2 years
  PFS means from the first use of the investigational product until disease progression or death, whichever occurs first, the disease progression will be evaluated by the investigator according to RECIST1.1 and iRECIST standards.
Investigator-assessed duration of remission(DoR). (Phase 1b) | 2 years
  DoR is defined as the time from the first CR or PR assessment by the investigator according to the RECIST1.1 and iRECIST criteria to tumor progression or death from any cause, whichever occurs first.
Investigator-assessed disease control rate (DCR). (Phase 1b) | 2 years
  It is defined as the percentage of the sum of CR, PR and disease stable for at least 4 weeks (SD≥4 weeks) evaluated by the investigator according to the RECIST1.1 and iRECIST standards.
Investigator-assessed overall survival (OS) and 1-year OS rate.(Phase 1b) | 2 years
  OS defined as the time from the first use of the investigational product to death from any cause. 1-year OS rate defined as the proportion of subjects surviving within 1 year after the first dose.
Investigator-assessed objective response rate (ORR). (Phase II) | 2 years
  ORR refers to the percentage of subjects with confirmed CR or PR according to RECIST1.1 and iRECIST.
Investigator-assessed progression-free survival (PFS) . (Phase II) | 2 years
  PFS means from the first use of the investigational product until disease progression or death, whichever occurs first, the disease progression will be evaluated by the investigator according to RECIST1.1 and iRECIST standards.
Investigator-assessed duration of remission(DoR). (Phase II) | 2 years
  DoR is defined as the time from the first CR or PR assessment by the investigator according to the RECIST1.1 and iRECIST criteria to tumor progression or death from any cause, whichever occurs first.
Investigator-assessed disease control rate (DCR). (Phase II) | 2 years
  It is defined as the percentage of the sum of CR, PR and disease stable for at least 4 weeks (SD≥4 weeks) evaluated by the investigator according to the RECIST1.1 and iRECIST standards.
Investigator-assessed overall survival (OS) and 1 year OS rate. (Phase II) | 2 years
  OS defined as the time from the first use of the investigational product to death from any cause. -year OS rate defined as the proportion of subjects surviving within 1 year after the first dose.
The type, frequency, severity and outcome of adverse events (TEAE) and serious adverse events (SAE) that occurred during the treatment period. (Phase II) | 2 years
  The toxicity was evaluated according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) (version 5.0) Grade.
Number of prticipants with abnormal laboratory values and/or Adverse Events that are related to treatment. (Phase II) | 2 years
  The laboratory values include 1. Routine blood test: Including complete blood count with differential. 2.Routine urine test: including specific gravity, pH, urine glucose, protein, ketone bodies and blood cell. 3.Serum biochemistry: Including ALT, AST, ALP, TP, ALB, TBIL, DBIL, GLU, BUN/UREA, Cr, K+, Na+, Cl-, Ca2+, P, TG, TC, HDL, LDL, and AMY/LIP. 4.Coagulation function: Including at least international normalized ratio (INR), activated partial thromboplastin time (APTT), fibrinogen (FIB), thrombin time (TT); if the international normalized ratio (INR) is not available, replace it with prothrombin time (PT). 5.Thyroid function test includes: serum thyroid stimulating hormone (TSH), free triiodothyronine (FT3), and free thyroxine (FT4); if FT3 and FT4 are not available, replace them with T3 and T4. 6.Troponin I or troponin T content: only during the screening period and when clinical indications (such as cardiac events occur).
Number of participants with abnormal vital signs values and/or Adverse Events that are related to treatment.(Phase II) | 2 years
  The vital signs include body temperature, heart rate, and respiratory frequency and blood pressure.
Number of participants with abnormal ECG and echocardiography values /or Adverse Events that are related to treatment.(Phase II) | 2 years
  During the screening period, it is necessary to repeat the inspection three times before the first administration, with an interval of about 5 minutes between each time. Calculate the QTc interval and calculate the mean (corrected using Fridericia's formula). If the inspection time in the screening period is ≤ 7 days before the first administration, the review may not be necessary according to the judgment of the investigator. Check once a week in the 1st cycle of phase Ib, check once on the 1st and 15th days of the 2nd cycle, and check once every 3 weeks from the 3rd cycle. Use echocardiography or multi-gate angiography scan to check the left ventricular ejection fraction.
Number of participants with aphysical examination values /or Adverse Events that are related to treatment.(Phase II) | 2 years
  A full physical examination in the screening period and at the end-of-treatment visit, including head, eyes, ears, nose, throat, neck, heart, chest (including lungs), abdomen, four limbs, skin, lymph nodes, nervous system, and subject's general condition. Body height and body weight are measured at the first visit, and then body weight is measured at each of the subsequent visits. Targeted physical examination will be conducted at other visits by the investigator.
ORR in PD-L1 positive and negative populations. | 2 years
  Collect subjects' pathological sections for evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No